CLINICAL TRIAL: NCT05794360
Title: A Randomized Controlled Trial (RCT) of the Impact of School-based Sport Research Program on Children's Physical Activity, Executive Function, and Academic Achievement
Brief Title: ACtive Children Enhance LEaRning and AttenTION: A Randomized Controlled Trial (RCT)
Acronym: ACCELERATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00003226
Record Dates: First submitted 2022-12-07; First posted 2023-04-03 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-03

CONDITIONS: Physical Inactivity
Keywords: physical activity; school; cognition; academic performance; executive function
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Acceleration

STUDY DESIGN:
Intervention Model Description: 2 arm clustered RCT. Two levels of clustering: The students (level 1) will be clustered within the classroom (level 2).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACCELERATION (Experimental): Both study arms occurred during participants' PE class, once a week for 45 minutes for 10 weeks. The ACCELERATION curriculum is designed to improve children's MVPA through learning and practicing new and challenging sport skills in a fun and free-will learning environment that includes not only school but also home environment. The ACCELERATION focuses on introducing the ball to the child at a basic level. Ball mastery is a soccer term that simply refers to the ability to manipulate and play with the ball using all parts of the foot. Since this program was an individual pursuit, not a team endeavor, it was imperative that each student has their own ball during the PE class. The trained undergraduate interns assisted PE teachers to deliver this program to classrooms assigned into the treatment arm. The program trains parents via virtual workshops on delivering the program at home.
  Interventions: Behavioral: ACtive Children Enhance LEaRning and AttenTION (ACCELERATION)
- Standard PE (No Intervention): Classrooms assigned to the control group received a 45-minute weekly regular PE curriculum for 10 weeks designed to meet state-mandated requirements. For the same research school, a standard PE curriculum was also delivered by the same PE teacher who delivered the intervention curriculum. However, additional training and support were not provided to PE teachers for the implementation of a regular PE curriculum.

INTERVENTIONS:
Behavioral: ACtive Children Enhance LEaRning and AttenTION (ACCELERATION) — A diverse group of key informants (i.e., PE teachers, school athletic department director) and community stakeholders (i.e., professional soccer coaches, Houston Dynamo Academy director) were engaged to help the research team design, modify, and implement the ACCELERATION curriculum to ensure program relevance and appeal. There are several components that described below make our program design both comprehensive and highly adaptable for optimal reach and effectiveness. These include staff development training, parent workshops, on-site and virtual developmental programs, delivery and implementation support from community stakeholders, online resources, family engagement events, equipment donations to improve activity, and on-going support and mentoring services for parents and school-based educators.
  Arms: ACCELERATION

SUMMARY:
The goal of this clinical trial is to test the effectiveness of sport-based physical education (PE) curriculum on activity behaviors (moderate to vigorous physical activity and sedentary behavior), executive functions, and academic performance in elementary school-aged children, particularly among low-income ethnic minorities. The main questions it aims to answer are:

* Whether a school-based sport program can improve child engagement in school-time moderate-to-vigorous physical activity (MVPA) and total daily MVPA, compared to a control group (standard PE class)?
* Whether a school-based sport program can improve child executive functions and academic performance, compared to a control group (standard PE class)?

Participants randomized to receive the ACtive Children Enhance LEaRning and AttenTION (ACCELERATION) intervention (treatment) received

* 45-minute weekly for 10 weeks soccer (ball mastery exercises) curriculum led by trained PE teachers during the school PE lesson time.
* Homework required practicing learned ball mastery skills daily for 15-20 minutes at home. A required ball was provided to them.
* Virtual parent workshops, which required the attendance of parents of study participants to improve their understanding of all about the program

Researchers will compare the control group, who received a regular PE class curriculum, to see if there are any differences in child activity behaviors, executive functions, and academic performance.

ELIGIBILITY:
Inclusion Criteria:

1. Any student enrolled in 3rd or 4th-grade classes were eligible to participate in the study.
2. Participation in an extracurricular sports activity wasn't an exclusion criterion for this study.

Exclusion Criteria:

1. Students were excluded if they had serious physical (e.g., asthma, heart diseases), developmental (e.g., autism, attention-deficit hyperactivity), or learning (e.g., dyslexia, dyscalculia, dysgraphia) disorders that prevented them from participating in intervention activities
2. Students who participated in a physical activity intervention within the last 6 months were excluded.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 257 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Average Accelerometer-measured MVPA/day at 10 weeks | baseline and post (immediate after 10 weeks of the intervention)
  MVPA behaviors were assessed objectively with accelerometers (GT3X+ Actigraph, Pensacola, FL). Trained research staff instructed the students to wear the accelerometer on the right hip for 8 days, which allowed participant to adapt to wearing the device and to achieve the study goal of 2 valid wear days per child as consistent with school-based evaluations. A valid day were defined as ≥600 minutes wear time per day. Freedson's age specific cut points for children 6 to 18 years old will be used to determine the intensity of activity.

SECONDARY OUTCOMES:
Change from Baseline in the Average Accelerometer-measured Sedentary Time/day at 10 weeks | baseline and post (immediate after 10 weeks of the intervention)
  Sedentary behaviors were assessed objectively with accelerometers (GT3X+ Actigraph, Pensacola, FL). Trained research staff instructed the students to wear the accelerometer on the right hip for 8 days, which allowed participant to adapt to wearing the device and to achieve the study goal of 2 valid wear days per child as consistent with school-based evaluations. A valid day were defined as ≥600 minutes wear time per day. Freedson's age specific cut points for children 6 to 18 years old will be used to determine the intensity of activity.
Change from Baseline in the Mean Dimensional Change Card Sort Test Score at 10 weeks | baseline and post (immediate after 10 weeks of the intervention)
  NIH Toolbox (appropriate for ages 7+) iPad Cognitive Battery utilized to deliver Dimensional Change Card Sort Test. This task measured the cognitive flexibility of children. Children were shown an on-screen target image and instructed to select one of two images matching the target on either shape or color.
Change from Baseline in the Mean Flanker Inhibitory Control and Attention Test Score at 10 weeks | baseline and post (immediate after 10 weeks of the intervention)
  NIH Toolbox (appropriate for ages 7+) iPad Cognitive Battery utilized to deliver Flanker Inhibitory Control and Attention Test. For this task, children were shown an arrow flanked by two additional arrows on each side and instructed to choose an on-screen button matching the direction of the middle arrow.
Change from Baseline in the Mean Picture Sequence Memory Task Score at 10 weeks | baseline and post (immediate after 10 weeks of the intervention)
  NIH Toolbox (appropriate for ages 7+) iPad Cognitive Battery utilized to deliver Picture Sequence Memory Task. Children were shown a narrated sequence of images corresponding to common activities- "How to go to the Park", followed by images depicting children playing on swings, feeding ducks. The same sequence was repeated and the participant was asked to recall the proper sequence.
Change from Baseline in the Mean the State of Texas Assessments of Academic Readiness (STAAR) Standardized Test Scores at 10 weeks | baseline and post (immediate after 10 weeks of the intervention)
  This test emphasizes students' readiness for success in the grade that follows by assessing the knowledge attained in the current grade level. Students in 3rd and 4th grade are tested on the following subjects, reading, mathematics.

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Johnston, PhD, Principal Investigator — University of Houston
Locations (1):
- KIPP Houston Public Schools, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diamond A, Lee K. Interventions shown to aid executive function development in children 4 to 12 years old. Science. 2011 Aug 19;333(6045):959-64. doi: 10.1126/science.1204529. PMID 21852486
- [Background] Diamond A, Ling DS. Conclusions about interventions, programs, and approaches for improving executive functions that appear justified and those that, despite much hype, do not. Dev Cogn Neurosci. 2016 Apr;18:34-48. doi: 10.1016/j.dcn.2015.11.005. Epub 2015 Dec 7. PMID 26749076
- [Background] Eime RM, Young JA, Harvey JT, Charity MJ, Payne WR. A systematic review of the psychological and social benefits of participation in sport for children and adolescents: informing development of a conceptual model of health through sport. Int J Behav Nutr Phys Act. 2013 Aug 15;10:98. doi: 10.1186/1479-5868-10-98. PMID 23945179
- [Background] Basterfield L, Reilly JK, Pearce MS, Parkinson KN, Adamson AJ, Reilly JJ, Vella SA. Longitudinal associations between sports participation, body composition and physical activity from childhood to adolescence. J Sci Med Sport. 2015 Mar;18(2):178-82. doi: 10.1016/j.jsams.2014.03.005. Epub 2014 Mar 15. PMID 24704422